CLINICAL TRIAL: NCT01122381
Title: Pharmacologic and Genetic Evaluation of a C. Elegans Model for Migraine
Brief Title: Comparison of a Drug and Placebo in the Prevention of Migraine Headaches
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Thomas Jefferson University (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B5043-R
Record Dates: First submitted 2010-05-10; First posted 2010-05-13 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Headache, Migraine
Keywords: headache, migraine; depression; disability evaluation; weight gain
MeSH Terms: conditions — Migraine Disorders; Depression; Weight Gain | interventions — Ethosuximide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1-ethosuximide (Experimental): ethosuximide blinded capsules of 250mg ESX; titration up to 4 capsules qd (expected) or 5 or 6 capsules for efficacy (not to exceed "30mg"/kg/d) vs maximum tolerability
  Interventions: Drug: ethosuximide
- Arm 2-placebo comparator (Placebo Comparator): placebo same size blinded capsules as the 250mg ESX; similar titration up to 4 capsules qd (expected) or 5 or 6 capsules for efficacy (not to exceed "30mg"/kg/d) vs maximum tolerability
  Interventions: Other: placebo comparator

INTERVENTIONS:
Drug: ethosuximide — ethosuximide (ESX)
  Other Names: zarontin
  Arms: Arm 1-ethosuximide
Other: placebo comparator — placebo
  Arms: Arm 2-placebo comparator

SUMMARY:
The purpose of this study is to determine whether ethosuximide works better than placebo in the prevention of episodic migraine among veterans.

DETAILED DESCRIPTION:
Chronic and episodic headaches in veteran populations include migraine, transformed migraine, and post-traumatic headache with migrainous features. More and better prophylactic drugs with fewer side effects (such as weight gain) are needed to treat these disabling, refractory conditions which generally have less than a 50% response rate to preventative treatments.

Rare forms of severe familial hemiplegic migraine (FHM) are considered channelopathies and can be caused by mutations in a calcium channel gene. Serotonin is also known to be a critical neurotransmitter in migraine based on the pharmacology of acute and preventative treatments. We previously identified a "migraine" signaling pathway in an invertebrate C. elegans "hemiplegic migraine" model of a mutant calcium channel upstream from transforming growth factor-beta (TGF-beta) and showed that low serotonin levels can be rescued by treatment with the childhood antiepileptic drug ethosuximide (ESX).

Objective: We propose to test our findings from this invertebrate migraine model to determine its relevance to humans in the prevention of episodic migraine.

Primary Aim: Determine whether ethosuximide (ESX) will be significantly more effective than placebo in reducing migraine headache days. We propose a 3 year, double blind, phase 1/2 randomized, 2:1 ESX:placebo controlled parallel trial in episodic migraineurs comparing migraine headache days during the last 4 weeks of treatment to a pre-treatment 4 week baseline.

ELIGIBILITY:
Inclusion Criteria:

* Must be a veteran.
* The number of migraine days per 4-week period is to be 4-14 for a period of 3 months prior to screening for entry into the trial.
* Migraine must have been occurring for 6 months preceding entry into the trial and age of onset should be before age 60 years.
* Migraine must be at least moderate severity and interrupt daily activities in some respect at least 3 times per month.
* As long as the veteran can easily distinguish nonmigraine headaches from migraine, there is no limit on the number of non migraine headache days allowed. "Transformed migraine" headaches due to medication over usage will be excluded according to exclusion criteria #4.
* Migraine diagnosis:

Veterans with headache must have migraine categorized using the International Headache Society (I.H.S.) criteria as illustrated below for the two main types with and without aura.

Criteria for migraine without aura (I.H.S. 1.1)

* > 5 attacks
* headache lasting 4-72 hours when untreated or not successfully treated.
* headache with two of the following characteristics

  * unilateral,
  * pulsating,
  * moderate to severe intensity,
  * aggravation by exertion.
* one of the following occurs with headache

  * nausea and/or vomiting
  * photophobia and phonophobia

Criteria for migraine with aura (I.H.S. 1.2)

* at least 2 attacks
* at least three of the following characteristics:

  * One or more fully reversible aura symptoms indicating focal cerebral cortical - and/or brain stem dysfunction.

One or more aura symptoms of the following types:

* Homonymous visual disturbance
* Unilateral parenthesis and/or numbness
* Unilateral weakness
* Aphasia or unclassifiable speech difficulty

  * At least one aura symptom develops gradually over more than 4 minutes or, 2 or more symptoms occur in succession.
  * No aura symptom lasts more than 60 minutes. If more than one aura symptom is present, accepted duration is proportionally increased.
  * Headache follows aura with a free interval of less than 60 minutes. (It may also begin before or simultaneously with the aura). Headache, nausea and/or photophobia usually follow neurological aura symptoms directly or after a free interval of less than an hour. The headache usually lasts 4-72 hours, but may be completely absent (1.2.5, acephalgic migraine).

Exclusion Criteria:

* Veterans with migraine plus other systemic disorder will be excluded if migraine onset was temporally related to onset of the systemic disorder.
* Blood pressure elevations (must be < borderline values 135/85 for 4 weeks before enrollment into the study). Current treatment for hypertension with beta-blockers, calcium channel blockers, or ace inhibitors not allowed.
* Use of other prophylactic migraine drugs (requires a washout phase) and cannot have failed more than two other prophylactic drugs for migraine.
* Excessive use of acute pain medicines, including narcotics (>10 days month). Those using non-narcotics could be tapered off over 4-8 weeks.
* Receiving disability or seeking disability for headache or chronic pain.
* Significant neck pain or cervicogenic contributors to chronic headache.
* Significant depression, anxiety, post-traumatic stress disorder, or other disabling psychiatric condition.
* Known allergies or serious side effects with ESX or succinimides in the past.
* Known liver or significant renal disease.
* Women veterans of child-bearing age who do not have adequate birth control.
* Chronic bone marrow suppression.
* Using psychogenic or other sedating maintenance drugs.
* History of porphyria.
* History of cluster headache. 15.History of other CNS disease.
* Age younger than 18 years and greater than 65.
* Women veterans who are breastfeeding.
* Veterans with familial hemiplegic migraine (FHM).

Ongoing exclusions during the study:

* The addition of other migraine prophylactic headache medicines is not allowed. 2. New drugs cannot be added that aggravate headache (nitrates, dipyridamole, niacin).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy L Gardner, MD, Principal Investigator — VA Pittsburgh Health Care System
Locations (1):
- VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary Care and Neurology Clinic prescreening and recruitment from VA Pittsburgh hospitals during the following periods:
  1/14/11-4/1/11; 1/14/12-3/19/12; 2/4/13-3/12/14. Average prescreening of datawarehouse records for eligibility = 2954 subjects/month.
  Average prescreening electronic chart review for eligibility = 265 subjects/month.
Pre-assignment Details: 5 consented. Initial 4 week baseline period uses headache diary to confirm headache days prior to randomization. 3/5 enrollees did not begin baseline phase; 1 lost to f/u, 1 dis-enrolled due to study interruption, 1 dis-enrolled shortly after consent when another physician began a study excluded drug. 2 enrollees did complete baseline phase.
Groups:
- Arm 1-drug Treatment: migraineurs with 4-14 headache days per month that meet all inclusion/exclusion criteria
  ethosuximide: ethosuximide (ESX) 250mg blinded capsules; begin 250mg qd titrating up to 1000mg qd (expected) or 1250mg qd, or 1500mg qd /30mg/kg/d maximum for efficacy goal of < 50% reduction in headache days versus maximum tolerability
- Arm 2-placebo: migraineurs with 4-14 headache days per month that meet all inclusion/exclusion criteria
  placebo comparator: placebo same size blinded capsules as the 250mg ESX; similar titration up to 4 capsules qd (expected) or 5 or 6 capsules for efficacy (not to exceed 30mg/kg/d) vs maximum tolerability
Period: Overall Study
Arm/Group | Arm 1-drug Treatment | Arm 2-placebo
Started | 1 | 1
Completed | 1 (Subject never took the drug per review of ESX levels after unblinding) | 0
Not Completed | 0 | 1
Not completed — study terminated early | 0 | 1

BASELINE CHARACTERISTICS:
Population: Enrollees who completed baseline period and randomization.
Groups:
- Arm 1: migraineurs with 4-14 headache days per month that meet all inclusion/exclusion criteria
  ethosuximide: ethosuximide (ESX) 250mg blinded capsules; begin 250mg qd titrating up to 1000mg qd (expected) or 1250mg qd, or 1500mg qd /30mg/kg/d maximum for efficacy goal of < 50% reduction in headache days versus maximum tolerability
- Arm 2: placebo same size blinded capsules as the 250mg ESX; similar titration up to 4 capsules qd (expected) or 5 or 6 capsules for efficacy (not to exceed "30mg"/kg/d) vs maximum tolerability
  placebo comparator: placebo same size blinded capsules as the 250mg ESX; similar titration up to 4 capsules qd (expected) or 5 or 6 capsules for efficacy (not to exceed 30mg/kg/d) vs maximum tolerability
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Migraine Headache Days Per 4 Week Period Comparing the Last 4 Weeks of Treatment to a 4 Week Pre-treatment Baseline.
Description: Compare number of migraine headache days pre and post treatment between the ESX and placebo group.
  Study terminated early-no outcome data available. The single subject assigned to study drug did not actually take it according to subsequent review of ESX drug levels.
Time Frame: 4 weeks, end of treatment and pre-treatment baseline
Groups:
- Arm 1-ethosuximide: Study was terminated early-no outcome data available. Only one subject was assigned to study drug arm but did not actually take it according to subsequent review of ESX drug levels.
- Arm 2-placebo Comparator: Study was terminated early-no outcome data available. Only one subject was assigned to study placebo but was dis-enrolled after titration phase due to study termination.
Arm/Group | Arm 1-ethosuximide | Arm 2-placebo Comparator
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- Arm 1- Ethosuximide: ethosuximide blinded capsules of 250mg ESX; subject was titrated up to 4 capsules qd
- Arm 2- Placebo Comparator: placebo blinded capsules of "250mg"; subject was titrated up to 4 capsules qd
Arm/Group | Arm 1- Ethosuximide | Arm 2- Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1- Ethosuximide (N=1) | Arm 2- Placebo Comparator (N=1)
hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — grade 1, mild
fatigue (General disorders) | 1 (1) | 1 (1) — grade 1, mild
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — grade 1, mild
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — grade 1, mild
somnolence (Nervous system disorders) | 1 (1) | 0 (0) — grade 1, mild
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — grade 1, mild

LIMITATIONS AND CAVEATS:
Early termination occurred due to inadequate recruitment of episodic migraineurs in a population meeting too many exclusion criteria; resulting in no subjects available for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No